CLINICAL TRIAL: NCT03815773
Title: PRospective Multicenter Observational Study on Transfusion Practice in Vv-ECMO Patients: The PROTECMO Study
Acronym: PROTECMO
Status: Completed | Type: Observational
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Collaborators: Medical University of Vienna (Other); University of Maryland, College Park (Other); University of Milan (Other); University of Milano Bicocca (Other); Pitié-Salpêtrière Hospital (Other); Hospital Vall d'Hebron (Other); St Vincent's Hospital, Sydney (Other); Columbia University (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Hospital Sao Joao (Other); Azienda Policlinico Umberto I (Other); University of Bari (Other); University of Turin, Italy (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRRB/15/17
Record Dates: First submitted 2018-12-17; First posted 2019-01-24 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Transfusion Related Complication; Hemorrhage; Anticoagulant-induced Bleeding
Keywords: ECMO; PRBC; Fresh frozen Plasma; Fibrinogen; Antithrombin III; Bleeding; Anticoagulation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Over the past decade, the use of extracorporeal membrane oxygenation (ECMO) for respiratory support in adults has increased. Several trials have highlighted how red blood cells transfusion can cause several negative effects and, currently, a restrictive transfusion trigger in critically ill patients is widely accepted.

The optimal management of anticoagulation targets and transfusion practice in veno-venous-ECMO (VV-ECMO) patients is still under debate. Traditionally, the threshold for transfusions of packed red blood cells (PRBC) in ECMO is aimed at keeping hemoglobin (Hb) values in the normal range (12-14 g/dL), but some case series have shown how the Hb target can be lower, and with comparable clinical outcomes.

While there are extensive reviews on predicted ECMO survival, and management (even with many debated issues), there is a significant knowledge gap in understanding the benefits and risks of transfusions during VV-ECMO Methods/Design: Prospective observational multicenter study. The principal aim is to describe current effective blood product usage, during VV-ECMO. The secondary aim is to describe in a large cohort of ECMO patients the current anticoagulation strategy and bleeding episodes occurrence.

The study will be conducted at a multicenter level including in each center all consecutive adult vv-ECMO patients during one year up. The data collection will include pre-ECMO characteristics, transfusion strategies and blood test results during the first twenty-eight days after ECMO cannulation or until the end of ECMO support if the length is shorter, and clinical outcomes up to the end of ICU stay.

The descriptive variable end points for the primary aim will be the daily and the total amount of PRBC and other blood products (Plasma, Platelets, Fibrinogen, Antithrombin III).

The descriptive variable end points for the secondary aim will be the type and dose of anticoagulation, and episodes of bleeding according to site and severity.

Expected Results: A collaborative combination of ECMO centers will evaluate prospective data of transfusion practices during ECMO. The investigators would be able to describe the currently strategy for administration of blood products, anticoagulation and the effective incidence of bleeding episodes worldwide.

DETAILED DESCRIPTION:
Background Over the past decade, the use of extracorporeal Membrane Oxygnation (ECMO) for respiratory support in adults has vastly increased. Veno-venous ECMO (VV-ECMO) can be initiated in case of Acute Respiratory Distress Syndrome (ARDS) as salvage therapy for patients with profound gas exchange abnormalities despite protective lung ventilation and other rescue therapies. Many aspects of ECMO management are still under debate despite the increasing number of cases. Among these debated topics there is certainly the optimal management of transfusion practice.

Several trials have recognized how red blood cells transfusion can cause several negative effects, including transfusion related immune reactions, the potential transmission of diseases, the development of transfusion-related complications (such as transfusion-related acute lung injury - TRALI - or transfusion-associated circulatory overload - TACO) and immunosuppression. On the other hand, anemia can also cause a potential increase in morbidity and mortality in critically ill patients, and in ECMO is an even greater critical issue in reducing delivery of oxygen (DO2).

Moreover, despite improvement in technology and care, complications related to ECMO are still high, and frequently involve an imbalance in the coagulation status due to anticoagulant use in the presence of coagulopathy. Consequently, the risk of thrombosis (presumably microthrombosis) and hemorrhage remain to be high. In the case of ongoing bleeding, transfusion of Packed Red Blood Cell (PRBC) is required to support desired haemoglobin levels.

Traditionally, the threshold for PRBC transfusions in ECMO is aimed to maintain hemoglobin (Hb) values in the normal range (12-14 g/dL). Despite this, there is considerable uncertainty regarding the optimal haemoglobin threshold for the use of PRBC transfusions in anemic patients during ECMO support.

Prompted by the general reappraisal of PRBC transfusion use, some case series using lower target for Hb during vv-ECMO support have been published. However, such protocols do not use/suggest a definitive trigger/target of Hb.

There is also some evidence that a higher number of transfusions in ECMO patients is associated with worse outcomes. However, such a relationship is difficult to assess given the large number of factors influencing transfusion practice in this setting: target of anticoagulation, frequent bleeding episodes, the peculiar characteristics of the circuits that can cause mechanical damage, activation of inflammation, and consumption of platelet and coagulation factors, to name but a few.

Moreover, most of the available data on transfusions during ECMO are heterogeneous, usually including VV-ECMO and veno-arterial-ECMO (VA-ECMO) configuration, and mixing adults with neonatal and pediatric cohorts, which are historically more represented.

In this context, the decision of giving a transfusion during ECMO support is still a real challenge since several parameters have to be taken into account at the same time. A strict trigger has not yet been defined in this population, and the literature on critically ill patients suggests a relevant reduction in the amount of transfusion.

Rationale for the study Providing adequate DO2 can be approached in several ways during vv-ECMO support, but the hemoglobin target is always a critical point, and a relevant piece of the puzzle of assuring the best oxygenation in patients affected with acute respiratory failure (ARF). There may be important variations between hospitals and countries in the use of PRBC transfusions, which may impact patient outcome. Large scale, national, and international studies are currently lacking.

There is a significant knowledge gap in understanding the benefits and risks of transfusion during VV-ECMO.

An international multicenter study will evaluate prospective observational data of transfusion practices during VV-ECMO, analyzing it in light of anticoagulation and bleeding episodes.

Aim of the study The PROTECMO study is aimed at being a collaborative study including a large number of ECMO centers worldwide, describing, in real practice,

1. Incidence of major bleeding events and amount of blood product transfused
2. Type, trigger and level of anticoagulation adopted

Study Design: international multicenter prospective observational cohort study. For the primary outcome PRBC will be evaluated as total amount during the ECMO run and in the first 28 days also as daily amount. The total amount of PRBC, adjusted for the ECMO length of stay, will be evaluated in light of pre-ECMO parameters (age, comorbidities, postoperative state and severity scores) and of daily data (bleeding episodes, ECMO blood flow, dieresis, CRRT, Hb, major events). Daily occurrence of PRBC transfusion will be described according to pre-ECMO characteristics and daily parameters (Hb, bleeding, hemodynamics, renal function, circuit change).

Plasma, platelets, Fibrinogen, Antithrombin III administration will be evaluated according to pre-ECMO data and according to daily APTT level (or other coagulation monitoring adopted), bleeding episodes, sepsis occurred For the secondary outcomes type of anticoagulant will be described as well as daily dose and daily target for the parameter targeted (APTT, ACT, r-TEG, anti-Xa according to local protocol). Anticoagulation will be described in relation to pre-ECMO parameters and daily episodes of bleeding and occurrence of sepsis.

Bleeding episodes will be described according to site (airway - including tracheotomy - oro-nasal, gastric, intrathoracic, abdominal, intestinal, retroperitoneal, urinary tract, other) and classified according to severity following 5 adjusted categories of the Bleeding Academic Research Consortium (BARC) score: Type 0, no bleeding; Type 1, Any overt bleeding that requires heparin infusion rate reduction or PRBC transfusion (provided Hb drop was related to bleeding); Type 2, any overt bleeding that requires heparin infusion rate reduction and packed red blood cells transfusion or non-surgical procedure to stop bleeding (provided Hb drop was related to bleeding); Type 3, Any life-threatening bleeding that required PRBC transfusion and surgical intervention for control of bleeding or ECMO discontinuation; Type 4: any fatal bleeding.

Every patient included will be registered for baseline values, and will then be followed for ECMO management and transfusion management daily for the first 28 days or until ECMO weaning if the ECMO run will be shorter than the observation time. Daily parameters will be recorded. Moreover, data will be recorded for every PRBC, Plasma, Platelets transfusion event. The patients will be observed for the clinical outcomes until they are discharged from the ICU and 6-months mortality will be recorded. Considering that according the Extracorporeal Life Support Organization summary, the average length of respiratory ECMO run is about 12 days we believe that the majority of ECMO run will be fully covered by the observation period and, at least, it will be paradigmatic of a center's actual practice and, at the same time, will assure a considerable sample size of transfusion events.

Data will be reported according to the STROBE (Strengthening the reporting of observational studies in epidemiology) statement checklist.

Study conduction Given the explorative nature of this study, the required number of patients was not calculated, but considering at least 10 patients/year for each center (considered the worst prediction) we imagine that the included patients will be at least 100 in Italy and we presume to enroll at least a double number worldwide.

Study duration

* Transfusions decisions for each patient will be recorded daily for 28 days after ECMO cannulation or until the end of ECMO support if the length is < 28 days.
* Patients will be observed until ICU discharge with a follow up to sixth months for mortality
* The inclusion period will be 12 months for each center.

Data collection methods Data will be recorded using pre-printed CRF by the principal investigator (PI) in each center or directly they will be recorded online. All data will be reported in a centralized online and Web-based fully encrypted database (REDCAP)

Data will include clinical characteristics: baseline demographics, basic biological values (e.g., blood gas, hemoglobin), primary diagnosis, comorbidities, underlying etiology of acute respiratory failure, severity of illness (e.g., SOFA, SAPS 2), type of ECMO, and the size of the cannulas.

ECMO management data will be collected daily for 28 days. Additionally, fluid balance, adverse events, Hb and all hematological data, anticoagulation management and monitoring will be collected every 24 hours.

For 28 days, transfusion amounts and values of Hb, HTC, Platelets, will be recorded.

Bleeding will be evaluated according to site and severity according to 5 adjusted categories of the Bleeding Academic Research Consortium (BARC) score.

Data will also be collected for the duration of mechanical ventilation, duration of ECMO, and ICU length of stay. Clinical outcome assessment will be made, with date of death, ICU discharge, hospital discharge, sixth month mortality.

Statistical Analysis Descriptive statistics including frequency (percentage), median and interquartile range (IQR) will describe overall population and groups of survivors and non-survivors.

In order to describe current transfusion practice the amount of PRBC, Plasma and Platelets, will be described as units and ml and as a number of transfusions adjusted for ECMO length of stay and considering the concomitant bleeding episodes.

Fibrinogen and Antithrombin III will be described as mg or units respectively and as a number of administration.

Anticoagulation will be reported as type, mean dosage and the confidence interval (CI 95%).

Hb average level and the confidence interval (CI 95%) will be reported. Baseline categorical and continuous variables will be compared for transfusion and ECMO weaning groups. In particular categorical variables will be compared with chi-square tests and continuous variables will be compared with Student's T-test, or Wilcoxon rank-sum tests, otherwise.

Multiple COX regression analysis will be used in order to explore the impact of confounding factors such as baseline patient severity, ECMO length of stay, bleeding episodes and possible others covariates and factors that will be observed and raised relevance during the first exploratory or univariate analysis. The impact of relevant confounding factors such as length of ECMO run, pre-ECMO severity scores, pre-ECMO administration of transfusions will be analyzed separately and together in multiple analyses.

In particular daily RBC transfusion will be studied according to the association to renal function, fluid balance, worst Hb level, episodes of bleeding, use of vasopressors, ECMO blood flow.

A p-value less of than 0.05 will be considered significant. Data handling and analyses will be done with SAS 9.4 software (SAS Institute Inc, Cary, NC, USA) and R 3.3 software (R Foundation for Statistical Computing).

Ethics: Informed Consent and Treatment of personal data The study will be conducted in compliance with the current Helsinki Declaration and the standards of good clinical practice.

The study involves the enrollment of patients undergoing extracorporeal membrane oxygenation support and therefore unable to express a consent.

Every participating center will have to ask the permission to their Ethic Committee or other relevant and competent authorities according to the local rules.

At ISMETT, according the Italian rules (and we strongly suggest to follow the same at the other centers), the investigators will apply the following practice about informed consent as it was approved by the Ethic Committee. The participating centers will be supperted with approval by ISMETT Ethic Committee and providing materials and translated informed consent either for the participation in the study and for the data protection policy.

According to the art. 82 of the Codice Privacy the investigators will ask for a consent for the treatment of personal data of the patients that for the particular support of the ECMO are almost always sedated at least at the beginning of the ECMO run - so they have to be considered temporarily unable to express a consent - to those that have legal authority over them or to the immediate relatives or to a person cohabiting with them or - failing these - to the person in charge of the facility where the data subject is hosted. In case the patient is able to an informed consent it will be asked to himself.

In the case of following improvement of neurological condition of the patient we will ask for a consent directly to the patient as soon as we will consider him again able to express a valid consent.

The results of the research will be diffused as aggregate data and in ways that will not allow in any case the identification of the enrolled patients.

Safety The present study, giving its observational design, has a complete safety profile.

There will be no additional interventions or measurements other than those that are standard of care at the participating center. All clinical activity will follow the well established protocols for ECMO support at each participating center and consequently the patients are at no risk by in participating in the study.

Predefined subgroup analyses If the sample size will be adequate, as explorative analyses, some subgroup analyses will be performed according to the following predefined plan.

Exploratory analyses will stratify data for center workload (<10, 10-20, >20 ECMO run per year), according to geographical areas (we imagine a stratification among continents but we will verify if, giving the amount of data, will be reasonable a country stratification), and for pre-ECMO severity scores (Preserve score and Respscore) divided in quartiles.

Moreover, by the repeated measurements of hemoglobin and eventual transfusion event, for each center we will profile the actual and effective hemoglobin accepted as a trigger. The outcome weaning from ECMO and effective ICU discharge will be stratified also according to different hemoglobin values (<7, 7-10, >10, >12).

Another subgroups analysis will involve age, considered a major impacting factor in survival during ECMO. Patients will be divided in quartiles and patients > 60 years old will moreover evaluated.

Jehovah's witnesses and all patients refusing transfusions for personal reasons, as well as patients affected with hematological malignances will be analyzed separately.

Expected results, potential benefit of the study and publication program A collaborative combination of ECMO centers will evaluate prospective data of transfusion practices during ECMO. The investigators would be able to describe the currently strategy for administration of blood products, anticoagulation and the effective incidence of bleeding episodes worldwide.

ELIGIBILITY:
Inclusion criteria:

- All consecutive patients who receive veno-venous ECMO for respiratory causes. Of note, considering the observational design of our study, patients can be included in other studies concurrently (this will be noted on the CRF).

Exclusion criteria:

- Refusal to include expressed by the relatives when tha patient is unconscious or by the patient when he is recovered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is prospective and, consequently, in each center all consecutive VV-ECMO adult patients who are eligible according to inclusion and exclusion criteria should be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 656 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Descriptive data of PRBC transfusion in patients receiving VV-ECMO | Day 28 after ECMO start
  Packed Red Blood Cells Transfused, amount
Descriptive data of Platelets transfusion in patients receiving VV-ECMO | Day 28 after ECMO start
  Platelets, amount
Descriptive data of Plasma transfusion in patients receiving VV-ECMO | Day 28 after ECMO start
  Plasma, amount
Descriptive data of Fibrinogen administration in patients receiving VV-ECMO | Day 28 after ECMO start
  Fibrinogen, amount
Descriptive data of Antithrombin III administration in patients receiving VV-ECMO | Day 28 after ECMO start
  Antithrombin III, amount

SECONDARY OUTCOMES:
Descriptive data of anticoagulation practices in patients receiving VV-ECMO | daily for 28 days
  Type of anticoagulant adopted during ECMO
Descriptive data of anticoagulation practices in patients receiving VV-ECMO | daily for 28 days
  Dose of anticoagulant adopted during ECMO
Descriptive data of bleeding episodes in patients receiving VV-ECMO | daily for 28 days
  Episodes of bleeding according to site and severity
Correlate the amount of transfusions to clinical outcomes | Day 28 after ECMO start
  ECMO weaning, Yes/Not

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Arcadipane, MD, Study Director — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies; Gennaro Martucci, MD, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- Ismett, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03815773/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03815773/ICF_001.pdf